CLINICAL TRIAL: NCT04177290
Title: A Phase I PK Similarity Study of Two Sintilimab Products Produced by Different Processes in Advanced or Metastatic NSCLC Patients
Brief Title: A PK Similarity Study of Two Sintilimab Products Produced by Different Processes in Advanced or Metastatic NSCLC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308K101
Record Dates: First submitted 2019-11-14; First posted 2019-11-26 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sintilimab (M1b) 200mg (Experimental)
  Interventions: Drug: Sintilimab (M1b)
- sintilimab (approved) 200mg (Active Comparator)
  Interventions: Drug: Sintilimab (approved)

INTERVENTIONS:
Drug: Sintilimab (M1b) — Intravenous infusion
  Arms: sintilimab (M1b) 200mg
Drug: Sintilimab (approved) — Intravenous infusion
  Arms: sintilimab (approved) 200mg

SUMMARY:
this is a phase I study comparing PK similarity of sintilimab by different production process (approved versus M1b) in Chinese advanced or metastatic NSCLC patients who have failed or been intolerant to at least one prior line of standard treatment

ELIGIBILITY:
Inclusion criteria

1. Histologically or cytologically confirmed locally advanced, recurrent or metastatic NSCLC patients who have received or been intolerant to at least one prior line of standard treatment.
2. No EGFR mutation or ALK rearrangement.
3. ECOG PS score 0 or 1.
4. BMI ≥ 21.0kg/m2 and ≤ 26.0kg/m2
5. Body weight ≥ 60.0kg and ≤ 75.0kg.
6. Adequate organ function per protocol-defined criteria.

Exclusion criteria

1. Exposure to any anti-PD-1, PD-L1, PD-L2 antibodies.
2. Allergic to any component of sintilimab.
3. Active autoimmune diseases.
4. Clinically unstable central nervous system metastasis.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
PK is defined as AUC0-∞. | 28 days

SECONDARY OUTCOMES:
PK is defined as Cmax. | 28 days
Safety of sintilimab (approved) versus sintilimab (M1b). AE is defined as treatment-related adverse events assessed by CTCAE v5.0. | from randomization through 90 days after last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, China